CLINICAL TRIAL: NCT06046508
Title: Migraine With Aura and Causal or Incidental Patent Foramen Ovale (PFO): Identification of Biomarker(s) to Select Patients Who Would Most Benefit From PFO Closure. The MANET Study
Brief Title: Migraine With Aura and Patent Foramen Ovale: Identification of Biomarkers to Select Patients In Whom Intervention Would Be Beneficial (MANET)
Acronym: MANET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: IRCCS Policlinico S. Donato (Other); Università di Cagliari (Unknown); Federico II University (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1934
Record Dates: First submitted 2023-08-21; First posted 2023-09-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-09

CONDITIONS: Migraine Headache; PFO - Patent Foramen Ovale
Keywords: platelets; prothrombotic platelets phenotype; metabolomics
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples will be used for platelet and erythrocyte function analysis and assessment of endothelial function
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sigle arm study: Patients with migraine headache with aura (MHA), patent foramen ovale (PFO) and previous neurological event (transient ischemic attack -TIA- or stroke) with clinical indication for percutaneous correction of the defect according to guidelines will be enrolled
  Interventions: Other: blood samples collection

INTERVENTIONS:
Other: blood samples collection — patients, who meet all the inclusion criteria and none of the exclusion criteria, will be enrolled and they will perform a blood withdrawal before PFO correction and 180 days after the intervention

SUMMARY:
This is a multicenter prospective observational study aimed to asses whether a specific prothrombotic platelet phenotype can discern migraine patients with PFO (patent forame ovale) - related symptoms from patients with incidental PFO. The study will also explore additional distinguishing features of causal and incidental PFO using a metabolomics approach. It involves the enrollment of well-characterized patient cohorts and an ex vivo approach using comparative cell biology models that reproduce the most critical aspects of the clinical scenario.

DETAILED DESCRIPTION:
Patients with PFO, who meet all the inclusion and none of the exclusion criteria, will be enrolled in the study. Patients will undergo percutaneous correction of PFO and the following evaluations as clinical practice:

* thrombophilic screening (factor V and II and MTHFR gene mutation); sampling for homocysteine, Protein C (Prot C), Protein S (Prot S) and antithrombin III assay;
* anatomic evaluation of the SIA (Saccular intracranial aneurysm) by color-doppler TT echocardiogram and intracardiac ultrasound for definition of the anatomy of the fossa ovalis: tunneled appearance; absence of SIA aneurysm; bulging of the SIA; convex right/left SIA aneurysm;
* quantification of right-left intracardiac shunt by CT doppler;
* classification of migraine according to Anzola scale at baseline visit, post PFO correction, at follow-up at 6 and 12 months.

For the purpose of the study, blood sampling will be performed for evaluation of platelet reactivity; oxidative stress, aggregability, and deformability of red blood cells; and isolation of Endothelial Colony Forming Cells (ECFCs) for analysis of endothelial function. The latter in particular will be evaluated in comparison with the endothelial function of 30 subjects without known disease with age > 18 years, enrolled as a control group.

All analyses will be performed before PFO correction and 180 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* presence of PFO with right-left shunt at baseline > 10 MES and during Valsalva > 20 MES
* previous Stroke or TIA
* positive MRI for ischemic outcomes
* SIA aneurysm or residual Chiari/Eustachian valve network
* thrombophilic screening positivity (MTHFR/prot C/prot S)
* cability to sign informed consent for study participation and adherence to planned clinical follow-ups

Exclusion Criteria:

* paroxysmal/refractory atrial fibrillation
* TSA vasculopathy
* left ventricular ejection fraction <30%
* moderate/severe mitral valve regurgitation
* need for long-term anticoagulant therapy
* allergy or intolerance to antiplatelet therapy
* nickel allergy
* severe chronic kidney disease (GFR < 30 mL/min)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MHA, PFO and previous neurological event (TIA or stroke) with clinical indication for percutaneous correction of the defect according to guidelines.
  As a control group, 30 subjects without known disease with age > 18 years will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of migraineurs patients with Platelet activation | through study completion, an average of 2 years
  Fresh whole blood will be stained for tissue factor (TF) expression, platelet activation markers [P-selectin and activated glycoprotein IIbIIIa] and annexinV binding to phosphatidylserine (PS). Flow cytometry analysis will be performed on fixed samples. Platelet procoagulant potential will be assessed by thrombin generation assay. The CAT assay (Chloramphenico Acetyltransferase) lwill be performed in the presence of a neutralizing anti-Tisse Factor (aTF) antibody (Ab) to assess the contribution of TF, and by adding an excess of exogenous phospholipids.
Number of migraineurs patients with high Thrombin generation levels | through study completion, an average of 2 years
  Flow cytometry MV characterization will be performed on stored patients' plasma samples. On the same plasma samples, MV procoagulant potential will be assessed by thrombin generation assay.
levels of the oxidative status in PFO patients | through study completion, an average of 2 years
  RBC (red blood cells) deformability and aggregability, generation of oxygen radicals in RBC and platelets of the overall enrolled population will be analyzed at T0 and at T1. Systemic redox status will be quantified by evaluating concentrations of both reduced glutathione (GSH) and its oxidized form GSSG (oxidized glutathione) on stored samples.
Number of migraineurs patients with Untargeted metabolomics | through study completion, an average of 2 years
  The metabolomic patterns of plasma, urine and platelets/ECFC (endothelial-colony forming cells) of the enrolled population will be investigated by a combined use of spectroscopy and multivariate and univariate statistical tools in order to identify the molecular fingerprint that could build a score able to identify patients with incidental PFO.

SECONDARY OUTCOMES:
Elucidate whether mechanical stress related to the right-to-left shunt may influence Erythrocyte behavior affecting in turn oxidative stress status | through study completion, an average of 2 years
  This will be accomplished ex vivo by using a microfluidic platform that recapitulates the specific shear stress profiles to which blood is exposed as it flows through the PFO
Assess whether a unique endothelial dysfunction profile identifies migraineurs with incidental PFO | through study completition, an average of 2 years
  Functional profiling will be carried out, by measuring proliferation, migration and in vitro angiogenesis. The pro-inflammatory and pro-thrombotic phenotype of the cells will be assessed using a panel of molecular markers. Platelet adhesion will be determined on resting and activated ECFC under flow conditions; thrombin generation will be measured using a cell-based assay.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Trabattoni, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (3):
- Italy (3):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan
  - Università di Cagliari, Cagliari
  - Azienda Ospedaliera Universitaria "Federico II", Napoli